CLINICAL TRIAL: NCT04597762
Title: Effect of Ciclosporin Eyedrops on Ocular Symptoms and Optical Quality in Patients With Sjögren Syndrome
Brief Title: Effect of Ciclosporin Eyedrops on Sjögren Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Hietzing (Other)
Responsible Party: Principal Investigator, Prof. Dr. Pia Vécsei-Marlovits, Pro. Dr. Pia Vécsei-Marlovits, Hospital Hietzing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SiccaIkervis
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Hydrocortisone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- right eye: Ciclosporin, left eye: Ciclosporin + Hydrocortisone (Experimental): Patients receive treatment with Ciclosporin eyedrops for the right eye and Ciclosporin eyedrops + Hydrocortisone eyedrops for the left eye
  Interventions: Drug: Cyclosporin; Drug: Hydrocortisone
- left eye: Ciclosporin, right eye: Ciclosporin + Hydrocortisone (Experimental): Patients receive treatment with Ciclosporin eyedrops for the left eye and Ciclosporin eyedrops + Hydrocortisone eyedrops for the right eye
  Interventions: Drug: Cyclosporin; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Cyclosporin — Cyclosporin eyedrops
Drug: Hydrocortisone — Hydrocortisone eyedrops

SUMMARY:
Keratoconjunctivitis sicca, also known as dry eye syndrome, is one of the most common ophthalmological diseases and is treated with tear substitutes to moisten the surface of the eye and, in more severe cases of this disease, with local anti-inflammatory therapy with corticosteroids or ciclosporin A. In patients with rheumatological diseases, such as Sjögren's syndrome, dry eye syndrome of severe extent occurs particularly frequently, which is why topical anti-inflammatory therapy is often necessary in these patients.

Aim of this study is to evaluate the treatment of severe dry eye syndrome with topical cyclosporin eyedrops with and without topical corticosteroids at the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe keratoconjunctivitis sicca defined by:
* Staining of the cornea ≥ grade III according to the Oxford scale
* OSDI value ≥ 12
* Age between 18 and 90 years
* Primary or secondary Sjogren's syndrome (defined according to the American-European Consensus Group criteria) with a stable course and unchanged treatment for 6 months

Exclusion criteria:

* Pregnancy (excluded with a pregnancy test in patients of childbearing potential)
* Children and young people up to the age of 18
* Eye surgery in the past 6 months
* Simultaneous participation in another study
* Regular use of eye drops, with the exception of tear substitutes
* Use of eye drops containing ciclosporin or glucocorticoids in the last 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
tearfilm breakup time | 6 months
  tearfilm breakup time measured with Fluorescein
corneal fluorescein staining | 6 months
  corneal fluorescein staining staged with Oxford grading scale, ranging from 0 (no staining) to 5 (maximal staining)
corneal optical aberrations | 6 months
  corneal optical aberrations measured with iTrace aberrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Augenabteilung - Klinik Hietzing, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No